CLINICAL TRIAL: NCT01931111
Title: Correlation Between Cardiovascular Risk Factors, Sedentary Behaviors and Maximal Oxygen Uptake in an Elderly Norwegian Population
Brief Title: Cardiovascular Risk Factors, Maximal Oxygen Uptake and Sedentariness: an Observational Study
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Gen100sub3
Record Dates: First submitted 2013-07-19; First posted 2013-08-29 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Aging
Keywords: physical activity; maximal oxygen uptake
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Norwegian Elderly Population

SUMMARY:
This is a substudy of the Generation-100 study (NCT01666340). The aim of this study is to find critical values for (1) maximal oxygen uptake and (2) sedentary behavior, below which cardiovascular risk parameter clustering is apparent in an elderly Norwegian population.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk at least 1km,
* born in 1938,1939,1940,1941 or 1942
* Sufficiently good health to be able to take part in the study, as determined by the researchers

Exclusion Criteria:

* Illness or disability that precludes exercise or hinders completion of the study
* Uncontrolled hypertension
* Symptomatic valve disease, hyper tropic cardio-myopathy or unstable angina
* Active cancer
* Test results indicating that study participation is unsafe
* Inclusion in other studies conflicting with participation in this one

Ages: 70 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly, norwegian
Sampling Method: Non-Probability Sample
Enrollment: 874 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
HDL blood correlation to maximal oxygen uptake | baseline
  Maximal oxygen uptake test on the bike or treadmill
LDL blood correlation to maximal oxygen uptake | baseline
C-reactive protein (CRP) correlation to maximal oxygen uptake | baseline

SECONDARY OUTCOMES:
sedentariness correlation with maximal oxygen uptake | baseline

CONTACTS AND LOCATIONS:
Overall Officials: dorthe stensvold, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zisko N, Nauman J, Sandbakk SB, Aspvik NP, Salvesen O, Carlsen T, Viken H, Ingebrigtsen JE, Wisloff U, Stensvold D. Absolute and relative accelerometer thresholds for determining the association between physical activity and metabolic syndrome in the older adults: The Generation-100 study. BMC Geriatr. 2017 May 16;17(1):109. doi: 10.1186/s12877-017-0497-1. PMID 28511695